CLINICAL TRIAL: NCT01866683
Title: Effects of Yoga on Heart Rate Variability, Electroencephalography, Quality of Life and Salivary Cortisol of Healthy Adult Subjets
Brief Title: Yoga Effects on Heart Rate Variability and Electroencephalography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Danilo Forghieri Santaella, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 184.583
Record Dates: First submitted 2013-05-23; First posted 2013-05-31 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Health Behavior; Quality of Life
Keywords: Yoga; Electroencephalography; Heart rate variability; Breathing Exercises; Quality of life
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): 1 month respiratory training
  Interventions: Behavioral: 1 month respiratory training; Behavioral: 1 month waiting period
- Group 2 (Experimental): 1 month waiting period
  Interventions: Behavioral: 1 month respiratory training; Behavioral: 1 month waiting period

INTERVENTIONS:
Behavioral: 1 month respiratory training — Bhastrika yoga respiratory training: 30 kapalabhati and 1 surya bedhana form 1 bhastrika
Behavioral: 1 month waiting period — waiting or detraining period

SUMMARY:
Since yoga breathing exercises are traditionally used to tranquilize the mind, and have a well-known positive effect on the cardiovascular system, it is our hypothesis that a respiratory yoga exercise named bhastrika pranayama may have positive effects on heart rate variability, electroencephalography, quality of life and salivary cortisol (stress hormone).

DETAILED DESCRIPTION:
The effects of yoga interventions on heart rate variability have been previously shown in our laboratory, having its efficacy in improving autonomic heart modulation of hypertensives and elderly subjets proven. However, there is a lack of data addressing the effects of such interventions on EEG patterns of health fit male subjects, as well as there are no study investigating if there is a relationship between heart autonomic modulation changes and EEG patterns. Thus, the aim of this study was to investigate the effects of 1 month respiratory yoga training on heart rate variability, EEG, salivary cortisol and quality of life of health fit male subjets.

ELIGIBILITY:
Inclusion Criteria:

* Young adults;
* Physically fit (engaged in physical activity at least 2-3 times a week);
* Non athletes;
* Possibility to follow protocol agenda.

Exclusion Criteria:

* Epileptic events in previous 5 years;
* Chronic allergic rhinitis, with airway occlusion;
* Oral bronchodilator usage;
* Beta blocker user;
* Any diagnosed cardiac rhythm alteration at rest;
* Cerebral dysrhythmia;
* Previous training in respiratory yoga exercises.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline electroencephalography measures of brain waves at 1 and 2 months | baseline, one month, two months
  64 active electrodes electroencephalography

SECONDARY OUTCOMES:
frequency domain heart rate variability | study entry, one month, two months
  R-R interval autoregressive spectral analysis
salivary cortisol | study entry, one month, two months
quality of life | study entry, one month, two months
  quality of life will be addressed by the World Health Organization Questionaire of Quality of Life in its brief form

CONTACTS AND LOCATIONS:
Overall Officials: Danilo F Santaella, Ph.D., Principal Investigator — University of São Paulo and Federal University of Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte - UFRN, Natal, Rio Grande do Norte, Brazil